CLINICAL TRIAL: NCT04159922
Title: Study of the Psychological Profile of Type 2 Diabetic Patients With Foot Wounds, Compared to Diabetic Patients Without Foot Wounds
Acronym: Bortner Pied
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VERGES 2019
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Foot Wound
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Foot Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetic patients with foot wounds
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Bortner self questionnaire: 14 items Cohen PSS Perceived Stress scale: 10 items quality of life scale: 32 items depression scale: 14 items

SUMMARY:
Several studies have highlighted the value of analyzing a patient's psychological profile with the Bortner scale questionnaire (defined as type A or B personality). This analysis helps to better understand and anticipate patients' behaviour, stress and compliance with their disease and its progression. The Type A personality profile combines hyperactivity, competitiveness and exaggerated ambition, while the B profile is characterized by lower sensitivity to stress and reduced competitiveness.

It has been shown that the type B psychological profile in patients with type 2 diabetes is an independent risk factor for inflammation and that, in type 1 diabetes, the type A psychological profile is associated with a decrease in the expression of the pro-inflammatory cFos gene.

Thus, the psychological profile appears to have an impact not only on the patient's behaviour but also on his or her biology.

It has never been determined whether the type A or B psychological profile assessed by Bortner's self-administered questionnaire can influence the development of foot wounds in patients with type 2 diabetes who often have a medically unfavourable prognosis and socio-economic difficulties. We would therefore like to study the psychological profile of these individuals in order to make comparisons with the data obtained in a previous study that included patients with type 2 diabetes who did not have a foot wound.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes
* patient > 18 years old
* with a diabetic foot wound
* person who has expressed non-opposiyion to participation in the study

Exclusion Criteria:

* a person who is not affiliated to national health insurance
* person subject to legal protection (curatorship, guardianship)
* person under limited judicial protection
* pregnant, parturient or breastfeeding woman
* adult unable to consent
* minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with type 2 diabetes with foot wounds
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Score of the Bortner self-questionnaire | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Verges B, Brands R, Fourmont C, Petit JM, Simoneau I, Rouland A, Legris P, Bouillet B, Chauvet-Gelinier JC. Fewer Type A personality traits in type 2 diabetes patients with diabetic foot ulcer. Diabetes Metab. 2021 Nov;47(6):101245. doi: 10.1016/j.diabet.2021.101245. Epub 2021 Mar 12. PMID 33722768